CLINICAL TRIAL: NCT02648828
Title: Understanding Physician Signout Risk Perception
Acronym: UPS
Status: Completed | Type: Observational
Sponsor: University of Pittsburgh (Other)
Collaborators: Carnegie Mellon University (Other)
Responsible Party: Principal Investigator, Janel Hanmer, Assistant Professor, University of Pittsburgh
Other Study IDs: PRO15040582
Record Dates: First submitted 2015-07-20; First posted 2016-01-07 (Estimated); Last update posted 2017-08-28 (Actual); Status verified 2017-08

CONDITIONS: Physician Judgment
Keywords: Judgment; risk assessment; clinical deterioration; cardiac arrest; Rothman Index
MeSH Terms: conditions — Clinical Deterioration; Heart Arrest

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Intern: Interns are in their first year of residency.
  Interventions: Other: Clinical deterioration
- Residents: Residents are in their 2nd or 3rd year of residency.
  Interventions: Other: Clinical deterioration
- Attendings: Attendings are physicians who have completed their residency.
  Interventions: Other: Clinical deterioration

INTERVENTIONS:
Other: Clinical deterioration — Patients at risk of clinical deterioration

SUMMARY:
The purpose of the study is to compare the ability of physicians and a statistical index (the Rothman score) to predict clinical deterioration over the next 24 hours. Clinical deterioration is defined as concern in change in vital signs or patient status requiring a call to the rapid response team, cardiopulmonary arrest, or transfer to the ICU.

DETAILED DESCRIPTION:
The proposed study will ask interns, residents, and attending physicians from general internal medicine teaching teams in a large teaching hospital to make predictions about the probability of their patient having a clinical deterioration in the next 24 hours. The investigators will compare these judgments to the Rothman index.

ELIGIBILITY:
Inclusion Criteria:

* Interns, residents, attendings in the Department of Medicine, Division of General Internal Medicine, University of Pittsburgh.
* Rotating on the general medical service at the University of Pittsburgh Medical Center - Presbyterian Hospital.

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Cohorts will be selected from the teaching teams of the University of Pittsburgh's General Internal Medicine wards.
Sampling Method: Non-Probability Sample
Enrollment: 132 (Actual)
Dates: Start 2015-07; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Difference between physician prediction of risk of clinical deterioration and Rothman Index | Six months
  Physicians will make judgments about the probability of clinical deterioration for each of their patients on a 0 (definitely won't) to 100 (certainly will) scale. Clinical deterioration is defined as rapid response, cardiopulmonary arrest, or ICU transfer in the next 24 hours. The Rothman Index is an index that predicts clinical deterioration. The area under the receiver operating curve (AUROC) will be calculated for physicians and the Rothman Index. The AUROC measures the association between the physician's judgment or Rothman Index and actual clinical deterioration. The AUROC of these two measures will then be statistically compared.

CONTACTS AND LOCATIONS:
Overall Officials: Janel A Hanmer, M.D., Principal Investigator — University of Pittsburgh; Deepika Mohan, MD, Principal Investigator — University of Pittsburgh; Alex Davis, PhD, Principal Investigator — Carnegie Mellon University
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Derived] Arnold J, Davis A, Fischhoff B, Yecies E, Grace J, Klobuka A, Mohan D, Hanmer J. Comparing the predictive ability of a commercial artificial intelligence early warning system with physician judgement for clinical deterioration in hospitalised general internal medicine patients: a prospective observational study. BMJ Open. 2019 Oct 10;9(10):e032187. doi: 10.1136/bmjopen-2019-032187. PMID 31601602